CLINICAL TRIAL: NCT02243800
Title: Study of the Efficacy and Safety of Cholecalciferol Supplementation on the Activity of Rheumatoid Arthritis in Patients With Vitamin D Deficiency
Acronym: SCORPION
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: CRINEX Laboratory (Unknown); BP 337 - 3 rue de Gentilly (Unknown); 92541 MONTROUGE Cedex FRANCE (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CHU-0205
Record Dates: First submitted 2014-09-16; First posted 2014-09-18 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Rheumatoid Arthritis; Vitamin D Deficiency
Keywords: Vitamin D; Rheumatoid arthritis; Cholecalciferol
MeSH Terms: conditions — Arthritis, Rheumatoid; Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- cholecalciferol (Experimental): One group will receive the study treatment: cholecalciferol One group will receive placebo
  Interventions: Other: cholecalciferol versus placebo
- placebo (Placebo Comparator): One group will receive the study treatment: cholecalciferol One group will receive placebo
  Interventions: Other: cholecalciferol versus placebo

INTERVENTIONS:
Other: cholecalciferol versus placebo

SUMMARY:
Vitamin D plays a key role in the regulation of calcium metabolism and bone physiology and also presents immunomodulatory effects. In contrast to healthy individuals, macrophages and synoviocytes synovium of patients with rheumatoid arthritis (RA) have receptors for vitamin D. In vitro, 1,25 Vitamin D inhibits T cell proliferation and cytokine synthesis and decreases pro-inflammatory process. There is an inverse relationship, at least in some epidemiological studies, between the circulating levels of 25OH vitamin D and the occurrence and / or activity of RA. The hypothesis of our study is that natural vitamin D supplementation in patients with RA and a vitamin D deficiency (vitamin D <30 ng / mL) improves functional disability.

DETAILED DESCRIPTION:
This is an interventional, multicenter (13 rheumatology units) randomized, double-blinded study against placebo, lasting 24 weeks. The main objective is to demonstrate that treatment with cholecalciferol improves functional disability (HAQ) in patients with RA not in remission (DAS28 VS> 2.6 and the investigator does not think to change the treatment in the 3 months after enrolment) and vitamin D deficiency (vitamin D <30 ng / ml). Secondary objectives will be to examine whether there is a decrease in disease activity (tender joint count, swollen joint count, VAS, EVA activity, ESR, CRP, EULAR criteria, ACR), a decrease in fatigue (FACIT EVA - fatigue), improved quality of life (SF36, EMIR, PASS, MOS) and the impact of RA (RAID).

ELIGIBILITY:
Inclusion Criteria:

- Patients with RA (ACR 1987) not in remission (DAS28> 2.6) in whom no change in treatment is considered by the investigator for at least 3 months, DMARD stable RA for at least 3 months and lack of infiltration in the last 2 months

- Serum 25-OH vitamin D <30 ng / ml

Exclusion Criteria:

* Arthritis resulting in class IV functional disability (according to the ACR criteria)
* Hypercalcemia (serum calcium> 2.6 mmol/L) and/or known hypercalciuria (calcium excretion> 4 mg / kg / day), history of renal colic, thiazideic therapy.
* Known hypersensitivity to vitamin D
* Patient refused to sign the consent form, pregnant or nursing women, patients minor, major patients under protection of the Act

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2011-11; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
The change in functional disability measured by the HAQ between the treated group and the placebo group. | at day 1

SECONDARY OUTCOMES:
The EULAR response criteria | at day 1
ACR response criteria | at day 1
The number of tender joints | at day 1
The number of swollen joints | at day 1
VAS pain | at day 1
EVA activity | at day 1
Parameters of inflammation | at day 1
Asthenia collected by VAS and FACIT - tiredness | at day 1
The impact of RA activity (RAID) | at day 1
Quality of life (SF-36, EMIR, MOS, PASS) | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Martin SOUBRIER, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France